CLINICAL TRIAL: NCT03527771
Title: Video-assisted Telephone CPR With the EmergencyEye-Software - a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, PD Dr. med. Wolfgang A. Wetsch, Principal Investigator, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EmergencyEye-POP
Record Dates: First submitted 2018-05-03; First posted 2018-05-17 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- unassisted CPR (No Intervention): unassisted CPR
- T-CPR (Active Comparator): telephone assisted CPR according to ERC Guidelines 2015
  Interventions: Drug: telephone-assisted CPR
- V-CPR (Experimental): video-assisted CPR according to ERC Guidelines 2015
  Interventions: Device: Video-assisted CPR

INTERVENTIONS:
Device: Video-assisted CPR — Emergency call using a Software capable of video Transmission for Video assistance in CPR
  Arms: V-CPR
Drug: telephone-assisted CPR — Emergency call with telephone assistance in CPR
  Arms: T-CPR

SUMMARY:
Technical advance as broad-bandwidth wireless internet coverage and the ubiquity utilization of smartphones has opened up new possibilities which surpass the normal audio-only telephony. High quality and real-time video-telephony is now feasible. However until now this technology hasn't been deployed in the emergency respond service.

In the hope of helping the detection of the cardiac arrest, offer the possibility to evaluate and correct via a video-instructed CPR (V-CPR) and to facilitate a fast localization of the emergency site, a new software (EmergencyEye®/RAMSES®) was developed which enables the dispatcher a video-telephony with the callers mobile terminal (smartphone) if suitable.

This technology hasn't been tested in a randomized controlled trail yet and no data exists that shows if V-CPR in comparison to T-CPR and non-instructed CPR leads to a better bystander CPR-performance.

DETAILED DESCRIPTION:
Technical advance as broad-bandwidth wireless internet coverage and the ubiquity utilization of smartphones has opened up new possibilities which surpass the normal audio-only telephony. High quality and real-time video-telephony is now feasible. However until now this technology hasn't been deployed in the emergency respond service.

In the hope of helping the detection of the cardiac arrest, offer the possibility to evaluate and correct via a video-instructed CPR (V-CPR) and to facilitate a fast localization of the emergency site, a new software (EmergencyEye®/RAMSES®) was developed which enables the dispatcher a video-telephony with the callers mobile terminal (smartphone) if suitable.

This technology hasn't been tested in a randomized controlled trail yet and no data exists that shows if V-CPR in comparison to T-CPR and non-instructed CPR leads to a better bystander CPR-performance.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer

Exclusion Criteria:

* healthcare providers (medical practitioners, nurses, paramedics etc.)
* pregnant women
* people with cardio-pulmonary and musculoskeletal diseases or any other impairment that would risk harm for the volunteer while performing CPR for 8 minutes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
CPR Compression Frequency | 8 minutes
  CPR Compression Frequency

SECONDARY OUTCOMES:
Compression Depth | 8 minutes
  Compression Depth
Cumulative No-Flow Time | Up to 8 minutes
  Cumulative No-Flow Time
Time to diagnosis | Up to 8 minutes
  Time to diagnosis
Time to beginning of chest compressions | Up to 8 minutes
  Time to beginning of chest compressions

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Intensive Care Medicine, University Hospital of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ecker H, Lindacher F, Adams N, Hamacher S, Wingen S, Schier R, Bottiger BW, Wetsch WA. Video-assisted cardiopulmonary resuscitation via smartphone improves quality of resuscitation: A randomised controlled simulation trial. Eur J Anaesthesiol. 2020 Apr;37(4):294-302. doi: 10.1097/EJA.0000000000001177. PMID 32073408